CLINICAL TRIAL: NCT00798850
Title: Randomised Controlled Trial of Percutaneous Transluminal Angioplasty (PTA) Versus a Supervised Exercise Programme (SEP) in the Management of Intermittent Claudication (IC) Due to Femoro-popliteal Disease
Brief Title: Trial of Nonsurgical Treatment of Intermittent Claudication Due to Femoro-popliteal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEY- REF-2424
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Femoropopliteal Disease; Intermittent Claudication
Keywords: Claudication; Vascular claudication; Peripheral Vascular Disease; Peripheral arterial disease; Peripheral arterial occlusive disease; Angioplasty; Femoral angioplasty; Superficial femoral artery; Femoral arterial disease; Exercise; Supervised exercise; Exercise therapy; Exercise programme; Infrainuginal; Quality of life; SF36; Questionnaire; VascuQol; Randomised; Randomised trial; Combination therapy; Intermittent Claudication due to Femoropopliteal Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1; Motor Activity | interventions — Angioplasty; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PTA (Active Comparator)
  Interventions: Procedure: Percutaneous Transluminal Angioplasty (PTA)
- SEP (Active Comparator)
  Interventions: Procedure: Supervised Exercise Programme (SEP)
- PTA+SEP (Active Comparator)
  Interventions: Procedure: Combined Treatment

INTERVENTIONS:
Procedure: Percutaneous Transluminal Angioplasty (PTA) — PTA will be performed by a consultant interventional radiologist with no deviation from the standard protocol at Hull & East Yorshire Yospitals NHS Trust.
  Arms: PTA
Procedure: Supervised Exercise Programme (SEP) — SEP: Conducted 3 times per week for 12 weeks.The session will be supervised by a physiotherapist and conducted in the cardiac gym.
  Each session begins with gentle warming up exercises followed by an exercise circuit of 6 stations(2 minutes each).
  1. Station 1-Step-ups(20-cm high step,alternating leg after 10 step-ups)
  2. Station 2-Exercise bicycles
  3. Station 3-Knee extensions with weights(2kg beanbag)
  4. Station 4-Heel raises
  5. Station 5-Knee bends(Alternating legs after 10 bends)
  6. Station 6-Rest station(2Kg Biceps curls) Gentle walk for 2minutes in between the stations to recover.For first 6weeks patients complete one full circuit, followed by on extra station/week, thus by 12weeks patients will complete 2 full circuits.Finally patients perform a series of gentle stretching and cooling down exercises.
  This exercise programme was designed to comply with suggested guidelines based on a meta-analysis assessing the effectiveness of SEP for claudicants.
  Arms: SEP
Procedure: Combined Treatment — PTA will be performed according to routine protocol followed by enrollment of patient in SEP. SEP will commence in the week following PTA.
  Arms: PTA+SEP

SUMMARY:
Intermittent Claudication (IC)is a common condition characterised by pain in the muscles of the legs on exertion caused by "hardening of the arteries" and a reduced blood supply. The investigators know that the vast majority of people suffering from this condition remain stable and do not deteriorate, and thus in general the viability of legs is not at risk. The main aim of treatment, therefore, is to try and improve walking thus reducing the impact this problem has on patients life style. There are many methods of management of intermittent claudication, but the investigators do not know which produces the best results. This study aims to compare the short and medium term outcomes of exercise programmes, percutaneous transluminal angioplasty and a combination of the two treatments for patients with intermittent claudication.

DETAILED DESCRIPTION:
Intermittent claudication (IC) is a common problem in the UK's elderly population with a prevalence of 5 -10%. Intermittent claudication infers significant quality of life limitations, however, it is a disease which generally runs a benign course with >80% of patients remaining stable. Yet the annual mortality rate in claudicants approaches 5%, three times that of age and sex matched population, due to the high prevalence of co-morbidity. IC is under-recognised as a risk factor for coronary and cerebrovascular events. Sixty percent of claudicants die from coronary heart disease and 10% of them die from stroke. Treating the patient with claudication, therefore, is likely to pay high dividends in terms of reducing deaths from myocardial infarction and stroke. The most appropriate management of IC, therefore remains a topic for debate but potentially beneficial therapies include: supervised exercise programmes (SEP); & percutaneous transluminal angioplasty (PTA).

A recent Cochrane review of PTA versus non-surgical management for intermittent claudication highlighted only two appropriate studies. More recently the results of a randomized control trial from Sweden have been published. This emphasizes the dearth of reliable scientific data in this area. It is believed that aorta-iliac atherosclerosis is often a solitary disease as opposed to femoro-popliteal disease which is often a manifestation of more generalized atherosclerosis. Further, the 5-year PTA patency rates for aorta-iliac disease are much better than those for femoro-popliteal PTA. Therefore, PTA is a well-established treatment modality for aorta-iliac disease but its role in femoro-popliteal disease is debatable11. This trial aims to prove the most effective treatment modality for claudication due to femoro-popliteal disease.

The two treatment modalities in question work by different mechanisms. PTA increases the blood flow to the limb. Whereas, exercise works by a combination of factors including optimized structural and metabolic performance of skeletal muscle, improvement in rheological parameters, development of collaterals, improved walking technique and marked psychological benefit. Still the efficacy of any treatment modality in claudication is judged by improvements in the standard measures of lower limb ischaemia as suggested by the International Society of Cardiovascular Surgery (ISCVS). These are essentially segmental pressure measurements and walking distances.

The primary aim of any treatment for patients with peripheral vascular disease is to improve the quality of life (QoL) rather than prolong survival. Several studies have shown that the traditional measures of lower limb ischaemia bear little correlation to the patient's QoL and these therefore need to be assessed independently. Further, generic QoL measures on their own are not sensitive enough to detect minor changes in QoL and so disease-specific measures need to be included in the outcomes.

Evidence is accumulating that each episode of exercise to the onset of claudication pain followed by rest may be considered as a low-grade ischaemia-reperfusion injury (IRI). Repeated episodes of IRI may have a cumulative effect leading to vascular endothelial damage and progression of atherosclerosis. This may explain the excess cardiovascular mortality seen in these patients16. Most experimental work measuring the biochemical markers of IRI is done following an episode of acute exercise. Few studies have shown the effect of an exercise -training programme on the biochemical markers of IRI. We intend to investigate this as a secondary component to the trial.

Heat shock proteins (hsp) are ubiquitous proteins found in the cells of all organisms. They are mainly classified according to their molecular weight. In addition to being constitutively expressed heat shock proteins can be induced by a number of stressors including heat, ischaemia and oxidative stress. Members of the hsp70 family are the most extensively studied group of stress proteins and they have been implicated in the prevention of ischaemia-reperfusion induced apoptosis, necrosis and oxidative injury in a variety of cell types including the cardiac myocyte18. Studies have shown hsp and their antibodies in the serum of normal individuals. Anti-hsp70 antibody levels in serum have been shown to be higher in vascular patients (IC, critical ischaemia and aortic aneurysms). Heat shock proteins have been detected in atherosclerotic lesions in higher concentrations. It is postulated that hsp play a key role in the autoimmune pathogenesis of atherosclerosis. Levels of anti-hsp antibodies are elevated in patients with carotid and coronary atherosclerosis and this correlates with the degree of atherosclerosis. Measuring anti-hsp antibodies in patients with IC undergoing exercise over a period of time may provide further valuable evidence on the role of heat shock proteins in atherosclerosis.

The secondary outcome measures of cost effectiveness analysis will interest health planners and clinicians as the health service has limited resources and 'value for money' has become increasingly important.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic unilateral Intermittent Claudication Femoro-popliteal lesion Angioplastiable lesion on duplex > 3 months on BMT

Exclusion Criteria:

* Critical ischaemia Incapacitating systemic disease Inability to tolerate treadmill testing Ischaemic changes on ECG during treadmill testing Ipsilateral surgery / PTA in previous 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2002-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Treadmill walking distances - Intermittent claudication distance(ICD),maximum walking distance(MWD) | Pretreatment, 1, 3, 6, 12, 36, & 60 months post treatment
Ankle brachial pressure indices(ABPI) measured at rest and post exercise | Pretreatment, 1, 3, 6, 12, 36, & 60 months post treatment

SECONDARY OUTCOMES:
Patient Reported Walking Distances (PRWD) | Pre-treatment, 1, 3, 6, 12, 36, & 60 months post treatment
Clinical outcomes(PTA patency,re-intervention rates, fatal&non-fatal events,amputation,mortality and ISCVS outcome) | Pre-treatment, 1, 3, 6, 12, 36, & 60 months post treatment
Health economic analyses | Pre-treatment, 1, 3, 6, 12, 36, & 60 months post treatment
Markers of ischaemia reperfusion | Pre-treatment, 1, 3, 6, 12, 36, & 60 months post treatment
Heat-shock proteins | Pre-treatment, 1, 3, 6, 12, 36, & 60 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter T McCollum, FRCS, Principal Investigator — Academic Vascular Surgery Unit, University of Hull
Locations (1):
- Academic Vascular Surgery Unit, Vascular Laboratory, Alderson House, Hull Royal Infirmary, Hull, East Riding Of Yorkshire, United Kingdom

REFERENCES:
- [Background] Fowkes FG, Housley E, Cawood EH, Macintyre CC, Ruckley CV, Prescott RJ. Edinburgh Artery Study: prevalence of asymptomatic and symptomatic peripheral arterial disease in the general population. Int J Epidemiol. 1991 Jun;20(2):384-92. doi: 10.1093/ije/20.2.384. PMID 1917239
- [Background] Chetter IC, Spark JI, Dolan P, Scott DJ, Kester RC. Quality of life analysis in patients with lower limb ischaemia: suggestions for European standardisation. Eur J Vasc Endovasc Surg. 1997 Jun;13(6):597-604. doi: 10.1016/s1078-5884(97)80070-6. PMID 9236714
- [Background] van der Heijden FH, Eikelboom BC, Banga JD, Mali WP. Management of superficial femoral artery occlusive disease. Br J Surg. 1993 Aug;80(8):959-63. doi: 10.1002/bjs.1800800806. PMID 8402088
- [Background] Leng GC, Lee AJ, Fowkes FG, Whiteman M, Dunbar J, Housley E, Ruckley CV. Incidence, natural history and cardiovascular events in symptomatic and asymptomatic peripheral arterial disease in the general population. Int J Epidemiol. 1996 Dec;25(6):1172-81. doi: 10.1093/ije/25.6.1172. PMID 9027521
- [Background] Smith GD, Shipley MJ, Rose G. Intermittent claudication, heart disease risk factors, and mortality. The Whitehall Study. Circulation. 1990 Dec;82(6):1925-31. doi: 10.1161/01.cir.82.6.1925. PMID 2242518
- [Background] Davies A. The practical management of claudication. BMJ. 2000 Oct 14;321(7266):911-2. doi: 10.1136/bmj.321.7266.911. No abstract available. PMID 11030662
- [Background] Phillips MJ, Cowan AR, Johnson CD. Intermittent claudication should not be treated by surgery. Ann R Coll Surg Engl. 1997 Jul;79(4):264-7. PMID 9244069
- [Background] Fowkes FG, Gillespie IN. Angioplasty (versus non surgical management) for intermittent claudication. Cochrane Database Syst Rev. 2000;(2):CD000017. doi: 10.1002/14651858.CD000017. PMID 10796469
- [Background] Gelin J, Jivegard L, Taft C, Karlsson J, Sullivan M, Dahllof AG, Sandstrom R, Arfvidsson B, Lundholm K. Treatment efficacy of intermittent claudication by surgical intervention, supervised physical exercise training compared to no treatment in unselected randomised patients I: one year results of functional and physiological improvements. Eur J Vasc Endovasc Surg. 2001 Aug;22(2):107-13. doi: 10.1053/ejvs.2001.1413. PMID 11472042
- [Background] Chetter IC, Spark JI, Kent PJ, Berridge DC, Scott DJ, Kester RC. Percutaneous transluminal angioplasty for intermittent claudication: evidence on which to base the medicine. Eur J Vasc Endovasc Surg. 1998 Dec;16(6):477-84. doi: 10.1016/s1078-5884(98)80237-2. PMID 9894486
- [Background] Ernst E. Exercise: the best therapy for intermittent claudication? Br J Hosp Med. 1992 Sep 16-Oct 6;48(6):303-4, 307. PMID 1422544
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Barletta G, Perna S, Sabba C, Catalano A, O'Boyle C, Brevetti G. Quality of life in patients with intermittent claudication: relationship with laboratory exercise performance. Vasc Med. 1996;1(1):3-7. doi: 10.1177/1358863X9600100102. PMID 9546911
- [Background] Garratt AM, Ruta DA, Abdalla MI, Buckingham JK, Russell IT. The SF36 health survey questionnaire: an outcome measure suitable for routine use within the NHS? BMJ. 1993 May 29;306(6890):1440-4. doi: 10.1136/bmj.306.6890.1440. PMID 8518640
- [Background] Tisi PV, Hulse M, Chulakadabba A, Gosling P, Shearman CP. Exercise training for intermittent claudication: does it adversely affect biochemical markers of the exercise-induced inflammatory response? Eur J Vasc Endovasc Surg. 1997 Nov;14(5):344-50. doi: 10.1016/s1078-5884(97)80283-3. PMID 9413374
- [Background] Whitley D, Goldberg SP, Jordan WD. Heat shock proteins: a review of the molecular chaperones. J Vasc Surg. 1999 Apr;29(4):748-51. doi: 10.1016/s0741-5214(99)70329-0. No abstract available. PMID 10194511
- [Background] Gallino A, Mahler F, Probst P, Nachbur B. Percutaneous transluminal angioplasty of the arteries of the lower limbs: a 5 year follow-up. Circulation. 1984 Oct;70(4):619-23. doi: 10.1161/01.cir.70.4.619. PMID 6236912
- [Background] Powers SK, LOCKE And M, Demirel HA. Exercise, heat shock proteins, and myocardial protection from I-R injury. Med Sci Sports Exerc. 2001 Mar;33(3):386-92. doi: 10.1097/00005768-200103000-00009. PMID 11252064
- [Background] Pockley AG, Shepherd J, Corton JM. Detection of heat shock protein 70 (Hsp70) and anti-Hsp70 antibodies in the serum of normal individuals. Immunol Invest. 1998 Dec;27(6):367-77. doi: 10.3109/08820139809022710. PMID 9845422
- [Background] Pockley AG, Bulmer J, Hanks BM, Wright BH. Identification of human heat shock protein 60 (Hsp60) and anti-Hsp60 antibodies in the peripheral circulation of normal individuals. Cell Stress Chaperones. 1999 Mar;4(1):29-35. doi: 10.1054/csac.1998.0121. PMID 10467106
- [Background] Chan YC, Shukla N, Abdus-Samee M, Berwanger CS, Stanford J, Singh M, Mansfield AO, Stansby G. Anti-heat-shock protein 70 kDa antibodies in vascular patients. Eur J Vasc Endovasc Surg. 1999 Nov;18(5):381-5. doi: 10.1053/ejvs.1999.0885. PMID 10610825
- [Background] Roma P, Catapano AL. Stress proteins and atherosclerosis. Atherosclerosis. 1996 Dec 20;127(2):147-54. doi: 10.1016/s0021-9150(96)05952-7. PMID 9125304
- [Background] Wick G. Atherosclerosis--an autoimmune disease due to an immune reaction against heat-shock protein 60. Herz. 2000 Mar;25(2):87-90. doi: 10.1007/pl00001957. PMID 10829245
- [Background] Xu Q, Kiechl S, Mayr M, Metzler B, Egger G, Oberhollenzer F, Willeit J, Wick G. Association of serum antibodies to heat-shock protein 65 with carotid atherosclerosis : clinical significance determined in a follow-up study. Circulation. 1999 Sep 14;100(11):1169-74. doi: 10.1161/01.cir.100.11.1169. PMID 10484536
- [Background] Zhu J, Quyyumi AA, Rott D, Csako G, Wu H, Halcox J, Epstein SE. Antibodies to human heat-shock protein 60 are associated with the presence and severity of coronary artery disease: evidence for an autoimmune component of atherogenesis. Circulation. 2001 Feb 27;103(8):1071-5. doi: 10.1161/01.cir.103.8.1071. PMID 11222468
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Patterson RB, Pinto B, Marcus B, Colucci A, Braun T, Roberts M. Value of a supervised exercise program for the therapy of arterial claudication. J Vasc Surg. 1997 Feb;25(2):312-8; discussion 318-9. doi: 10.1016/s0741-5214(97)70352-5. PMID 9052565
- [Result] Mazari FA, Gulati S, Rahman MN, Lee HL, Mehta TA, McCollum PT, Chetter IC. Early outcomes from a randomized, controlled trial of supervised exercise, angioplasty, and combined therapy in intermittent claudication. Ann Vasc Surg. 2010 Jan;24(1):69-79. doi: 10.1016/j.avsg.2009.07.005. Epub 2009 Sep 17. PMID 19762206
- [Result] Mazari FA, Carradice D, Rahman MN, Khan JA, Mockford K, Mehta T, McCollum PT, Chetter IC. An analysis of relationship between quality of life indices and clinical improvement following intervention in patients with intermittent claudication due to femoropopliteal disease. J Vasc Surg. 2010 Jul;52(1):77-84. doi: 10.1016/j.jvs.2010.01.085. Epub 2010 May 14. PMID 20471779
- [Result] Mazari FA, Khan JA, Carradice D, Samuel N, Abdul Rahman MN, Gulati S, Lee HL, Mehta TA, McCollum PT, Chetter IC. Randomized clinical trial of percutaneous transluminal angioplasty, supervised exercise and combined treatment for intermittent claudication due to femoropopliteal arterial disease. Br J Surg. 2012 Jan;99(1):39-48. doi: 10.1002/bjs.7710. Epub 2011 Oct 21. PMID 22021102
- [Result] Mazari FA, Khan JA, Carradice D, Samuel N, Gohil R, McCollum PT, Chetter IC. Economic analysis of a randomized trial of percutaneous angioplasty, supervised exercise or combined treatment for intermittent claudication due to femoropopliteal arterial disease. Br J Surg. 2013 Aug;100(9):1172-9. doi: 10.1002/bjs.9200. PMID 23842831
- [Derived] Mazari FA, Khan JA, Samuel N, Smith G, Carradice D, McCollum PC, Chetter IC. Long-term outcomes of a randomized clinical trial of supervised exercise, percutaneous transluminal angioplasty or combined treatment for patients with intermittent claudication due to femoropopliteal disease. Br J Surg. 2017 Jan;104(1):76-83. doi: 10.1002/bjs.10324. Epub 2016 Oct 20. PMID 27763685